CLINICAL TRIAL: NCT05809947
Title: Regulation of Human Tendon and Skeletal Muscle Protein Turnover Following Tissue Injury: Mechanisms Behind Regeneration and Injury Preventive Adaptations
Brief Title: Mechanisms of Tissue Repair After Muscle Injury and Tendon Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Grith Højfeldt, Principal investigator, postdoc, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BBH150
Record Dates: First submitted 2023-03-17; First posted 2023-04-12 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Muscle; Injury, Quadriceps (Thigh); Tendon Strain
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Growth hormone/somatropin (Experimental): Somatropin over two weeks (33.3 ug/kg/day in the first week, 50 ug/kg/day in the second week)
  Interventions: Other: Neuromuscular electrical stimulation
- Placebo (Placebo Comparator): Injections of placebo/saline over two weeks
  Interventions: Other: Neuromuscular electrical stimulation

INTERVENTIONS:
Other: Neuromuscular electrical stimulation — One bout of neuromuscular electrical stimulation in conjunction with forced lengthening contractions on one leg
  Other Names: Neuromuscular electrical stimulation using Theta 4 channel stimulator from Chattanooga. Coupled with forced eccentric contractions.

SUMMARY:
The study is a 5-week human study including 24 18-35 year old healthy men. Each participant will have muscle injury and tendon strain induced in one leg using neuromuscular electrical stimulation in conjunction with forced lengthening contractions. The investigators will monitor the recovery from injury/strain over a 4 week period, in which half of the subjects will receive growth hormone (somatropin) to stimulate the connective tissue synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men
* BMI between 18.5-30 kg/m^2

Exclusion Criteria:

* Smoking
* Regular strength training within the last 3 months
* Current or former use of anabolic steroids or growth hormone
* Use of corticosteroids in the last 3 months
* Use of blood thinning medication
* Use of medication which can affect muscle protein synthesis
* Current or former drug og alcohol abuse
* Knee pain
* Previous participation in studies using deuterated water or alanine tracers

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-01-03 (Actual)

PRIMARY OUTCOMES:
Effect of somatropin on muscle protein synthesis 14 days after injury | 14 days
  The difference in fractional synthesis rate in muscle proteins 14 days after injury with or without 14 days treatment with somatropin. Measured using deuterated water

SECONDARY OUTCOMES:
Muscle protein synthesis 7 days after injury | 7 days
  The difference in fractional synthesis rate in muscle proteins 7 days after injury vs control (no injury) with or without 7 days treatment with somatropin. Measured using deuterated water
Muscle protein synthesis 14 days after injury | 14 days
  The difference in fractional synthesis rate in muscle proteins 14 days after injury compared to control leg (no injury). Measured using deuterated water.
Muscle protein breakdown 14 days after injury | 14 days
  The difference in fractional synthesis rate in muscle proteins 14 days after injury vs. control (no injury) with or without 14 days treatment with somatropin. Measured using stable isotop labelled alanine.
Muscle protein breakdown 7 days after injury | 7 days
  The difference in fractional synthesis rate in muscle proteins 7 days after injury vs. control (no injury) with or without 7 days treatment with somatropin. Measured using stable isotop labelled alanine.
Muscle protein breakdown 28 days after injury | 28 days
  The difference in fractional synthesis rate in muscle proteins 28 days after injury vs. control (no injury) with or without 14 days treatment with somatropin. Measured using stable isotop labelled alanine.
Histochemical staining of muscle cross sections 7 days after injury | 7 days
  Number of satellite cells, fibroblasts and immune cells in injured vs. control tissue (no injury), with and without growth hormone. Measured using histochemical staining of muscle cross sections
Histochemical staining of muscle cross sections 14 days after injury | 14 days
  Number of satellite cells, fibroblasts and immune cells in injured vs. control tissue (no injury), with and without growth hormone. Measured using histochemical staining of muscle cross sections
Histochemical staining of muscle cross sections 28 days after injury | 28 days
  Number of satellite cells, fibroblasts and immune cells in injured vs. control tissue (no injury), with and without growth hormone. Measured using histochemical staining of muscle cross sections
The effect of somatropin on tendon tissue synthesis | 7 days
  The difference in fractional synthesis rate in tendon proteins after 7 days placebo/treatment with somatropin. Measured using deuterated water
Tendon tissue synthesis 7 days after strain | 7 days
  The difference in fractional synthesis rate in tendon proteins 7 days after strain compared to control leg (no strain). Measured using deuterated water
Tendon tissue synthesis 7 days after strain with/without somatropin | 7 days
  The difference in fractional synthesis rate in tendon proteins 7 days after strain compared to control leg (no strain) with or without somatropin. Measured using deuterated water
Isometric muscle force output 7 days following injury | 7 days
  The difference in isometric muscle force output 7 days after injury vs. control (no injury) with or without 7 days treatment with somatropin.
Isometric muscle force output 14 days following injury | 14 days
  The difference in isometric muscle force output 14 days after injury vs. control (no injury) with or without 14 days treatment with somatropin.
Isometric muscle force output 28 days following injury | 28 days
  The difference in isometric muscle force output 28 days after injury vs. control (no injury) with or without 14 days treatment with somatropin.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
The IPD will be made available upon individual request once the study is finalised and published.